CLINICAL TRIAL: NCT00886444
Title: Comparative Evaluation of Various CMR Pulse-Sequences for Macrophage Imaging Using Ferucarbotran as Molecular Contrast Agent in Human Myocardial Infarction
Brief Title: Comparative Evaluation of Various Combinable Magnetic Resonance (CMR) Pulse-sequences for Macrophage Imaging Using Ferucarbotran
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Responsible Party: Principal Investigator, Udo Sechtem, Prof. Dr. med. U. Sechtem, Division of Cardiology, Robert-Bosch-Krankenhaus, Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIMINI-1; RBK-143
Record Dates: First submitted 2009-04-20; First posted 2009-04-23 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Acute Myocardial Infarction
MeSH Terms: interventions — ferumoxides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ferucarbotran (Experimental)
  Interventions: Drug: Ferucarbotran (Resovist)

INTERVENTIONS:
Drug: Ferucarbotran (Resovist) — single time intravenous bolus injection of a contrast agent
  Other Names: Resovist

SUMMARY:
The aim of this study is to:

* clarify whether macrophage imaging using ferucarbotran is able to delineate the region of myocardial infarction as accurate as gadolinium-based necrosis/fibrosis imaging;
* identify possible differences in infarct imaging using ferucarbotran for macrophage imaging compared to necrosis/fibrosis imaging with gadolinium-based compounds; and
* evaluate which MRI pulse-sequences maximise sensitivity for macrophage imaging with ferucarbotran in the setting of acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* acute myocardial infarction (STEMI or NSTEMI)

Exclusion Criteria:

* contraindication to CMR or Magnevist® or Resovist®

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-03; Primary Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Extent of myocardial infarction (as demonstrated with gadolinium-based necrosis/ fibrosis imaging compared to macrophage imaging using ferucarbotran) | within 5 - 15 days after myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Udo Sechtem, MD, Study Director — Robert Bosch Medical Center
Locations (1):
- Robert-Bosch-Krankenhaus, Division of Cardiology, Stuttgart, Germany